CLINICAL TRIAL: NCT03895502
Title: Optimal Duration of Anticoagulation Therapy for Isolated Distal Deep Vein Thrombosis in Patients With Cancer Study
Acronym: ONCO DVT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y0019
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Venous Thrombosis; Neoplasms; Anticoagulant
Keywords: Venous Thrombosis; Neoplasms; Anticoagulant
MeSH Terms: conditions — Venous Thrombosis; Neoplasms | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-month Edoxaban (Experimental): Edoxaban for 12 months
  Interventions: Drug: 12-month Edoxaban
- 3-month Edoxaban (Active Comparator): Edoxaban for 3 months
  Interventions: Drug: 3-month Edoxaban

INTERVENTIONS:
Drug: 12-month Edoxaban — Prescription of Edoxaban for 12 months
  Arms: 12-month Edoxaban
Drug: 3-month Edoxaban — Prescription of Edoxaban for 3 months
  Arms: 3-month Edoxaban

SUMMARY:
The purpose of this study is to determine the optimal duration of anticoagulation therapy (3 months versus 12 months) with direct oral anticoagulant (edoxaban) for isolated distal deep vein thrombosis.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), including pulmonary embolism (PE) and deep vein thrombosis (DVT), is a major health problem in the world. There have been many clinical studies evaluating PE and/or proximal DVT, although data on isolated distal DVT (IDDVT) has been quite limited. However, IDDVT was reported to account for about half of all the diagnoses of DVT detected on ultrasound in daily clinical practice, and optimal management strategies for these patients are becoming clinically more relevant. The current American College of Chest Physicians (ACCP) guidelines suggest the same approach for IDDVT patients with cancer as proximal DVT patients with cancer. However, whether anticoagulation therapy should be continued indefinitely remains uncertain and the duration of treatment in these patients might vary widely in daily clinical practice. Recently, some observational studies reported that IDDVT patients with cancer have a high risk of VTE recurrence, suggesting the benefit of prolonged anticoagulation therapy. In this open-label, superiority trial, we will randomly assign IDDVT patients with active cancer to receive either edoxaban for 3 months (short DOAC group) or edoxaban for 12 months (long DOAC group).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly found isolated distal deep vein thrombosis
* Patients complicated with active cancer
* Patients who are scheduled to be treated by anticoagulation therapy.

Exclusion Criteria:

* Patients with anticoagulation therapy for the index event before 10 days of allocation.
* Patient under anticoagulation therapy for the purpose of other than the index event.
* Patients with thrombolysis therapy or IVC filter at the Index event.
* Patients with creatinine clearance less than 30 ml/min.
* Patients who are expected to have a life prognosis of 3 months or less.
* Patients with pulmonary embolism.
* Patients who are not appropriate for the participation of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic VTE recurrence event or VTE related death event | 12 months
  Symptomatic VTE recurrence event is defined as PE and/or DVT with symptoms accompanied by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy. VTE related death event is defined as death due to a documented PE (either an objective test prior to death of the subject or PE detected during autopsy) or unexplained death (i.e. death without a clear alternate cause and not a primary consequence of subject's underlying cancer.)

SECONDARY OUTCOMES:
Major bleeding event (ISTH criteria) | 12 months
  Major bleeding is defined as International Society of Thrombosis and Hemostasis (ISTH) major bleeding, which consisted of a reduction in the hemoglobin level by at least 2 g/dL, transfusion of at least 2 units of blood or symptomatic bleeding in a critical area or organ.
All-cause death | 12 months
Symptomatic VTE recurrence event | 12 months
  Symptomatic VTE recurrence event is defined as PE and/or DVT with symptoms accompanied by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy.
VTE related death event | 12 months
  VTE related death event is defined as death due to a documented PE (either an objective test prior to death of the subject or PE detected during autopsy) or unexplained death (i.e. death without a clear alternate cause and not a primary consequence of subject's underlying cancer.)
Clinically relevant non-major (CRNM) bleeding | 12 months
  A bleeding event will be classified as a clinically relevant non-major bleeding event if it is overt (i.e. is symptomatic or visualized by examination) not meeting the criteria for major bleeding, requires medical attention or is associated with discomfort for the subject such as pain, or impairment of activities of daily life.
Clinically relevant bleeding | 12 months
  Clinically relevant bleeding is defined as major or CRNM bleeding.
Bleeding related death event | 12 months
  Bleeding related death event is defined as a bleeding event directly led to death. Examples of fatal bleeding events are an intracranial hemorrhage that led to herniation of the brain and death within 24 hours, and a massive gastrointestinal hemorrhage that results in shock, hemodynamic collapse, and death.
Unsuspected recurrent DVT by follow-up ultrasound examinations | 12 months
  Unsuspected DVT by follow-up ultrasound examinations is a thrombus that is detected during follow-up ultrasound testing without suspicion of DVT.
Unsuspected recurrent VTE by any imaging examinations | 12 months
  Unsuspected recurrent VTE is defined as thrombi that are detected during imaging testing performed for other reasons (e.g., computed tomography (CT) for cancer staging) and not for suspicion of DVT or PE.
Change of serum D-dimer levels during follow-up period | 12 months
Any adverse outcomes during invasive procedures | 12 months
  Adverse outcomes include bleeding events, recurrent VTE events, all-cause deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine, Kyoto, Japan

REFERENCES:
- [Derived] Nishikawa T, Yamashita Y, Fujita M, Morimoto T, Muraoka N, Umetsu M, Nishimoto Y, Takada T, Ogihara Y, Ikeda N, Otsui K, Sueta D, Tsubata Y, Shoji M, Shikama A, Hosoi Y, Tanabe Y, Chatani R, Tsukahara K, Nakanishi N, Kim K, Ikeda S, Yasui T, Yamamoto H, Ono K, Kimura T; ONCO DVT Study Investigators. D-dimer after 3 months of anticoagulation therapy and outcomes in cancer-associated isolated distal deep vein thrombosis. Blood Vessel Thromb Hemost. 2025 Feb 24;2(2):100063. doi: 10.1016/j.bvth.2025.100063. eCollection 2025 May. PMID 40766276
- [Derived] Chatani R, Yamashita Y, Morimoto T, Muraoka N, Umetsu M, Nishimoto Y, Takada T, Ogihara Y, Nishikawa T, Ikeda N, Otsui K, Sueta D, Tsubata Y, Shoji M, Shikama A, Hosoi Y, Tanabe Y, Tsukahara K, Nakanishi N, Kim K, Ikeda S, Mushiake K, Kadota K, Ono K, Kimura T. Edoxaban for 12 vs. 3 months in cancer-associated isolated distal deep vein thrombosis according to different doses: insights from the ONCO DVT study. Eur Heart J Cardiovasc Pharmacother. 2024 Aug 14;10(5):422-431. doi: 10.1093/ehjcvp/pvae028. PMID 38650055
- [Derived] Yamashita Y, Morimoto T, Muraoka N, Oyakawa T, Umetsu M, Akamatsu D, Nishimoto Y, Sato Y, Takada T, Jujo K, Minami Y, Ogihara Y, Dohi K, Fujita M, Nishikawa T, Ikeda N, Hashimoto G, Otsui K, Mori K, Sueta D, Tsubata Y, Shoji M, Shikama A, Hosoi Y, Tanabe Y, Chatani R, Tsukahara K, Nakanishi N, Kim K, Ikeda S, Mo M, Yoshikawa Y, Kimura T; ONCO DVT Study Investigators. Edoxaban for 12 Months Versus 3 Months in Patients With Cancer With Isolated Distal Deep Vein Thrombosis (ONCO DVT Study): An Open-Label, Multicenter, Randomized Clinical Trial. Circulation. 2023 Nov 21;148(21):1665-1676. doi: 10.1161/CIRCULATIONAHA.123.066360. Epub 2023 Aug 28. PMID 37638968